CLINICAL TRIAL: NCT07269249
Title: Real-world Efficacy and Safety of Neoadjuvant Dostarlimab in Patients With dMMR/MSI-H Locally Advanced Rectal Cancer
Acronym: RW-NEDOS
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: RW-NEDOS
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
Keywords: dostarlimab; mismatch repair-deficient LARC; real-world; retrospective-prospective study; neoadjuvant setting
MeSH Terms: interventions — dostarlimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Stage II-III rectal cancer (LARC): patients with dMMR/MSI LARC treated with neoadjuvant dostarlimab
  Interventions: Drug: Dostarlimab

INTERVENTIONS:
Drug: Dostarlimab — Dostarlimab 500 mg iv every 3 weeks for 9 cycles

SUMMARY:
This is an observational, retrospective-prospective, multicentre trial enrolling all patients included in the AIFA monitoring registry of Dostarlimab for the indication in rectal cancer. The aims of the study are to describe the clinical outcomes and safety of patients with dMMR/MSI-H locally advanced rectal cancer (LARC) receiving neoadjuvant dostarlimab in the real-world setting.

DETAILED DESCRIPTION:
The primary objective is to describe the activity of neoadjuvant dostarlimab in terms of objective response rate (RECIST 1.1).

Secondary objectives are:

1. To describe the activity of neoadjuvant dostarlimab in terms of:

   * complete clinical response rate at 6 and 12 months
   * time to clinical complete response
   * duration of clinical complete response
   * near-complete clinical response rate at 6 and 12 months
   * duration of near-complete clinical response
   * duration of objective response
   * rate of surgery (total mesorectal excision or local excision)
   * pathological complete response rate
   * objective response rate (RECIST 1.1) assessed by central radiological review.
2. To describe the safety of neoadjuvant dostarlimab in terms of: Adverse events/SAE incidence and outcome, time and duration of toxicity according to CTCAE v5.0.
3. To descrive the efficacy of neoadjuvant dostarlimab in terms of: event free-survival (EFS), organ preservation at 3 years, time to ditance recurrence and overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age > 18 years
* Histologically confirmed stage II-III rectal cancer
* dMMR/MSI status assessed locally by Immunohistochemistry, next-generation sequencing or PCR

For the retrospective part of the study:

* At least one dose of neoadjuvant dostarlimab from November 2023 (i.e. within the period of AIFA dostarlimab monitoring registry activation for the indication in rectal cancer, which is reimbursed according to the Italian law 648/1996, GU n.252 as of 27/10/2023)
* Eligible deceased or unreachable patients will also be included to avoid selection biases, in respect of the article 110 bis, paragraph 4 of the Italian Privacy Code (a Data Protection Impact Assessment will be produced and published on the Sponsor website before study initiation, and patients explicitly unwilling before death will be not included).

For the prospective part of the study:

- Inclusion in the AIFA dostarlimab monitoring registry for the indication in rectal cancer, to receive dostarlimab according to the Italian law 648/1996, GU n.252 as of 27/10/2023

Exclusion Criteria:

* - Distant metastasis
* Major cognitive dysfunction or psychiatric disorders
* Any previous systemic or local treatment for rectal cancer
* Dostarlimab received within an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (any sex/gender) with dMMR/MSI-H locally advanced rectal cancer treated with dostarlimab are eligible for this study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | after 3 , 6 and 9 cycles of dostarlimab. Each cycle is 21 days. Up to 6 months
  Defined as the percentage of trial participants having a CR or PR, as per RECIST v1.1.

SECONDARY OUTCOMES:
duration of clinical complete response | up to to 12 months
  defined as the time from the first documented date of clinical complete response to the date of documented local tumor regrowth, disease recurrence, or last available follow-up, whichever occurs first.
near-complete clinical response rate | at 6 and 12 months up to 12 months
  absence of mass at digital rectal exam, small mucosal irregularity or superficial ulcer no more than 2 cm in diameter at endoscopic exam, and no metastatic nodes at MRI.
duration of near-complete clinical response | up to 12 months
  defined as the time from the first documented date of near-complete clinical response to the date of documented conversion to complete clinical response, local tumor regrowth, disease recurrence, or last available follow-up, whichever occurs first.
rate of surgery (total mesorectal excision or local excision) | at 6 months (at the end of neoadjuvant dostarlimab)
  defined as the proportion of patients who undergo surgical resection of the primary tumor, including either total mesorectal excision (TME) or local excision
pathological complete response rate | after surgery (at 6 months)
  defined as a Tumor Regression Grade (TRG) 1 according to Mandard modified scoring system.
objective response rate assessed by central radiological review | fter 3 , 6 and 9 cycles of dostarlimab. Each cycle is 21 days. Up to 6 months
  defined as the percentage of trial participants having a CR or PR, as per RECIST v1.1.
safety of neoadjuvant dostarlimab | at the end of each cycle of dostarlimab (every 21 days ) up to 6 months
  Adverse events/Serious adverse events incidence and grading according to NCI-CTCAE v. 5.0
Event-free survival | up to 12 months
  defined as the time between dostarlimab starting and disease recurrence (local or distant), or disease progression (radiological or clinical) or second primary colorectal malignancy, or death from any cause, whichever comes first.
Time to distant recurrence | up to 12 months
  defined as the time between dostarlimab starting and distant disease recurrence or progression. Patients who do not have a distant recurrence and are alive at the end of the study will be censored at the date of the last assessment visit.
Overall survival | up to 12 months
  defined as the time between dostarlimab starting and death from any cause. Patients alive at the end of the study will be censored at the date of the last follow-up contact.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carmela Piccirillo, MD, Principal Investigator — National Cancer Institute, IRCCS Fondazione G. Pascale
Locations (2):
- Italy (2):
  - ASL Napoli 1, Presidio Ospedaliero Ospedale del mare, Oncologia medica, Napoli
  - IRCCS Fondazione G. Pascale, Unità Operativa Complessa Oncologia Addominale, Napoli

IPD SHARING:
Plan to Share IPD: Yes